CLINICAL TRIAL: NCT01278238
Title: Hemodynamic Effect of Prophylactic Phenylephrine Versus Lower Limb Compression in Women During Caesarean Section Under Spinal Anaesthesia
Brief Title: Optimization of Hemodynamic Conditions During Caesarean Section Under Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anestesiavdelingen Baerum Sykehus (Other)
Responsible Party: Principal Investigator, Jana Christine Kuhn, Dr.med., Anestesiavdelingen Baerum Sykehus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-013025-42
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Caesarean Section
Keywords: Hypotension; Caesarean section; Spinal anaesthesia; Lower limb compression / wrapping; Phenylephrine
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phenylephrine (Active Comparator)
  Interventions: Drug: Phenylephrine
- Lower limb compression (Active Comparator)
  Interventions: Device: Lower limb compression
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Phenylephrine — Intravenous infusion Dosage 0,25 microgram/kg bodyweight as bolus, continuous infusion with 0,25 microgram/kg/min
  Arms: Phenylephrine
Device: Lower limb compression — Tight bandaging of lower extremity up to hips with compression bandages
  Arms: Lower limb compression
Other: Placebo — Neither phenylephrine nor lower limb bandaging
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine wether intravenous Phenylephrine, administered as start bolus and following continuous infusion (specific dosage per weight), or optimal lower limb bandaging is more effective in preventing hypotension during caesarean section under spinal anaesthesia in healthy women.

The hypothesis is that the Phenylephrine model is superior to lower limb compression in preventing hypotension.

ELIGIBILITY:
Inclusion Criteria:

Healthy women Elective caesarean section under spinal anaesthesia Informed consent Age 18-40 ASA 1-2 BMI 18-32 prior to pregnancy Height 160-180 cm

Exclusion Criteria:

Any form of disease or anomalities:

Heart or vascular disease Cerebrovascular disease Other somatic or psychiatric disease Hypertension or preeclampsia Contraindication against spinal anaesthesia Anomalities concerning pregnancy and foster

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Invasive arterial bloodpressure | Until end of operation, up to roughly 1 hour

SECONDARY OUTCOMES:
pH value from umbilical vessels of the newborn | straight after delivery
APGAR score of the newborn | 1 + 5 + 10 minutes after delivery
Need for rescue pressor (ephedrine, phenylephrine) | Until end of operation, roughly 1 hour
Cardiac Output | Until end of operation, roughly 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Jana Christine Kuhn, Dr.med., Principal Investigator — Bærum sykehus
Locations (1):
- Bærum Sykehus, Rud, Akershus, Norway